CLINICAL TRIAL: NCT06014827
Title: Phase II Trial of the Addition of Biologically Guided Radiation Therapy (BgRT) and Stereotactic Body Radiation Therapy (SBRT) to Tyrosine Kinase Inhibitor in Oligoprogressive Oncogenic Positive Non-Small Cell Lung Carcinoma
Brief Title: Biologically Guided Radiation Therapy (BgRT) and Stereotactic Body Radiation Therapy (SBRT) to Tyrosine Kinase Inhibitor in Oligoprogressive Oncogenic Positive Non-Small Cell Lung Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22624; NCI-2023-06041 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22624 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-08-21; First posted 2023-08-28 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Specimen Handling; osimertinib; Magnetic Resonance Spectroscopy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (BgRT/SBRT) (Experimental): Patients continue to receive osimertinib PO QD in the absence of unacceptable toxicity. Patients undergo BgRT/SBRT every other day for 5 treatments. Patients then continue to receive osimertinib and are monitored via imaging. If additional progression is found, patients may receive additional BgRT/SBRT therapy. Treatment continues in the absence of > 5 sites of progression, unacceptable toxicity, or the stopping of osimertinib for more than 4 weeks.
  Patients undergo CT scan or PET/CT scan and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Osimertinib; Procedure: Positron Emission Tomography; Radiation: Stereotactic Body Radiation Therapy; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT or PET/CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Osimertinib — Given PO
  Other Names: AZD-9291; AZD9291; Mereletinib; Tagrisso
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Radiation: Stereotactic Body Radiation Therapy — Undergo BgRT/SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
Other: Survey Administration — Ancillary study

SUMMARY:
This phase II trial tests how well biologically guided radiation therapy (BgRT) and stereotactic body radiation therapy (SBRT) with osimertinib works for the treatment of EGFR positive non-small cell lung carcinoma that has spread from where it first started (primary site) to a limited number of anatomic sites (oligoprogressive). BgRT is radiation that uses specialized imaging to during treatment to target the active tumor and direct radiation to tumors in order to kill and shrink tumor cells. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Osimertinib is in a class of medications called kinase inhibitors. It works by blocking the action of a protein called EGFR that signals cancer cells to multiply. This helps slow or stop the spread of tumor cells. Giving BgRT with SBRT and osimertinib may kill more tumor cells in patients with oligoprogressive EGFR positive non-small cell lung carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the percent of patients receiving benefit at 6 months from the addition of BgRT/SBRT to first line osimertinib in EGFR positive non-small cell lung cancer (NSCLC) patients with oligoprogressive disease (disease control rate [DCR]).

SECONDARY OBJECTIVES:

I. To evaluate the tolerability of adding BgRT/SBRT to first line osimertinib in EGFR positive NSCLC patients with oligoprogressive disease.

II. To estimate the overall survival when adding BgRT/SBRT to first line osimertinib in EGFR positive NSCLC patients with oligoprogressive disease.

III. To describe the effect on quality of life (QOL) when adding BgRT/SBRT to first line osimertinib in EGFR positive NSCLC patients with oligoprogressive disease.

IV. To describe the effect on quantified fludeoxyglucose F-18 (FDG) uptake changes when adding BgRT to first line osimertinib in EGFR positive NSCLC patients with oligoprogressive disease.

V. To estimate local and distant control rates when adding BgRT/SBRT to first line osimertinib in EGFR positive NSCLC patients with oligoprogressive disease.

VI. To estimate the extracranial progression free survival (PFS) when adding SBRT to first line osimertinib in EGFR positive NSCLC patients with oligoprogressive disease.

VII. To estimate the time to treatment failure (TTF) when adding BgRT/SBRT to first line osimertinib in EGFR positive NSCLC patients with oligoprogressive disease.

VII. To estimate percentage of patients needing salvage BgRT/SBRT when adding SBRT to first line osimertinib in EGFR positive NSCLC patients with oligoprogressive disease.

EXPLORATORY OBJECTIVES:

I. To identify potential predictors of outcome when adding BgRT/SBRT to first line osimertinib in EGFR positive NSCLC patients with oligoprogressive disease.

II. To describe the changes in circulating tumor deoxyribonucleic acid (ctDNA) levels when adding BgRT/SBRT to first line osimertinib in EGFR positive NSCLC patients with oligoprogressive disease.

OUTLINE:

Patients continue to receive osimertinib orally (PO) daily (QD) in the absence of unacceptable toxicity. Patients undergo BgRT/SBRT every other day for 5 treatments. Patients then continue to receive osimertinib and are monitored via imaging. If additional progression is found, patients may receive additional BgRT/SBRT therapy. Treatment continues in the absence of > 5 sites of progression, unacceptable toxicity, or the stopping of osimertinib for more than 4 weeks.

Patients undergo computed tomography (CT) scan or positron emission tomography(PET)/CT scan and blood sample collection throughout the study.

After completion of initial radiation therapy, patients follow up at 1 week, 3 months, 6 months and 12 months and then for an additional year.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Age: >= 18 years
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Histologically confirmed advanced non-small cell lung cancer (NSCLC)
* The tumor harbors 1 of the 2 common epidermal growth factor receptor (EGFR) mutations known to be associated with epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKI) sensitivity (Ex19del or L858R), either alone or in combination with other epidermal growth factor receptor (EGFR) mutations, which may include T790M.
* Disease progression in the metastatic setting on PET or CT imaging when receiving first line standard/approved single agent osimertinib after having had stable disease (per Response Evaluation Criteria in Solid Tumors [RECIST] version [v] 1.1 or PET Response Criteria in Solid Tumors [PERCIST] v 1.0) for more than 6 months
* Disease progression must be in the form of 1-5 extracranial sites (any number of metastatic sites at initial diagnosis will qualify). For progression of the primary and oligoprogressive site(s), the primary should be treated with curative/local control intent. The primary, if progressing is considered as 1 site. Maximum of 3 lesions per organ (i.e. patient with 4 oligoprogressive sites in the lung would be excluded). Each lesion will be considered as 1 "site" so 3 lesions in the lung for example will be considered 3 sites. Patients with prior metastases that have been treated with ablative therapies before their current line of systemic therapy are eligible. Patients with brain metastases can be included but brain metastases must be treated (asymptomatic and have had no requirement for steroid medication for 1 week prior to the first dose of study drug and have completed radiation 2 weeks prior to the first dose of study drug) prior to enrollment (brain metastases [mets] will not be counted as a site of progression)
* Lesion(s) must be amenable to SBRT as determined by the radiation oncologist. If a patient is unable to receive a minimum of 30 Gy in 5 fractions they will not qualify
* At least one lesion must be amenable to BgRT which includes either a lung or bone metastasis, greater than or equal to 2 cm, which can also receive a minimum of 30 Gy in 5 fractions
* No prior systemic therapy for advanced disease other than osimertinib
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 4 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
* Patients must be able to swallow and retain oral medications
* Life expectancy of at least 6 months

Exclusion Criteria:

* Chemotherapy, radiation therapy, biological therapy, immunotherapy within 21 days prior to day 1 of protocol therapy (6 weeks for nitrosoureas or mitomycin C). Exceptions to this exclusion are brain radiation (2 weeks) and osimertinib
* Strong CYP3A4 inducers/ inhibitors within 14 days prior to day 1 of protocol therapy
* Patients receiving class 1A or class III antiarrhythmic agents within 14 days prior to day 1 of protocol therapy
* Drugs known to prolong the corrected QT (QTc) interval
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Clinically significant uncontrolled illness
* Active infection requiring antibiotics bacterial, viral, or fungal infections, requiring systemic therapy
* Known history of immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection
* Prior malignancy other than carcinoma in situ of the cervix, or nonmelanoma skin cancer, unless that prior malignancy was diagnosed and definitively treated 5 or more years prior to study entry with no subsequent evidence of recurrence. Patients with a history of low grade (Gleason score =< 6 =Gleason group 1) localized prostate cancer will be eligible even if diagnosed less than 5 years prior to study entry. Other malignancies with low probability of recurrence may be allowed with primary investigator (PI) approval
* Females only: Pregnant or breastfeeding
* Any malabsorption condition
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Diagnosis of congenital long QT syndrome
* New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on electrocardiogram (ECG)
* Clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroid medication for 1 week prior to the first dose of study drug and have completed radiation 2 weeks prior to the first dose of study drug
* Patients with active interstitial lung disease (ILD) / pneumonitis or with a history of ILD/ pneumonitis requiring steroids
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-07-11 (Estimated); Study Completion 2026-07-11 (Estimated)

PRIMARY OUTCOMES:
Percent of patients on planned protocol treatment | At 6 months
  Patient counts and percentages will be provided.

SECONDARY OUTCOMES:
Rate of all grades and grade >= 3 adverse events at least possibly related to study therapy | Up to 2 years
  As measured by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Observed toxicities will be summarized, for all patients in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.
Overall survival | From the date of study enrollment to the date of death from any cause, up to 2 years
  Will be estimated using the product-limit method of Kaplan-Meier. Two-sided 95% confidence intervals will be computed.
Change in quality of life (QOL) | From baseline to 3 months post initial stereotactic body radiation therapy (SBRT)
  As measured by Functional Assessment of Cancer Therapy-General (FACT-G) v4. Repeated QOL assessments will be tabulated and graphically displayed to describe the changes of QOL outcomes over time.
Change in fludeoxyglucose (FDG) uptake | From baseline to completion of SBRT, up to 2 years
  As measured by metabolic tumor volume and total lesion glycolysis at each fraction. Will be analyzed using independent student's t-test to compare normal variables and non-parametric tests including Wilcoxon's signed-rank test for paired data will be used to compare non-normally distributed variables. Repeated measures analysis of variance (ANOVA) will be used to test for differences at more than one time point. Correlation between metabolic tumor volume, total lesion glycolysis and circulating tumor deoxyribonucleic acid (ctDNA) and time to treatment failure (as described above) as well as overall survival will be explored using univariate and multivariate Cox regression.
Ratio of patients achieving local control and distant control | Up to 2 years
First occurrence of disease progression | From study entry to first occurrence of disease progression, up to 2 years
  By Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) v1.0 or Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. A progressive event will occur when: more than five sites of progression based on PERCIST or RECIST, inability to receive more biologically guided radiation therapy (BgRT)/SBRT or osimertinib, physician decision to come off study or change therapy, patient withdrawal of consent or death will all be considered events. Will be estimated using the product-limit method of Kaplan-Meier.
Time to treatment failure | From study entry to treatment failure, up to 2 years
  Will be estimated using the product-limit method of Kaplan-Meier. For time to treatment failure, a progressive event will occur when: more than five sites of progression based on PERCIST or RECIST, inability to receive more BgRT/SBRT or osimertinib, physician decision to come off study or change therapy, patient withdrawal of consent or death will all be considered events.
Ratio of patients needing salvage BgRT/SBRT | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Arya Amini, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - Yale University, New Haven, Connecticut